CLINICAL TRIAL: NCT04369469
Title: A Phase 3 Open-label, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Intravenously Administered Ravulizumab Compared With Best Supportive Care in Patients With COVID-19 Severe Pneumonia, Acute Lung Injury, or Acute Respiratory Distress Syndrome
Brief Title: Efficacy and Safety Study of IV Ravulizumab in Patients With COVID-19 Severe Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Met futility bar at interim analysis
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-COV-305
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Severe Pneumonia; Acute Lung Injury; Acute Respiratory Distress Syndrome; Pneumonia, Viral
Keywords: acute lung injury; acute respiratory distress syndrome; antibodies, monoclonal, humanized; COVID-19; hospitalization; pneumonia; severe pneumonia; severe acute respiratory syndrome; severe acute respiratory syndrome coronavirus 2; randomized controlled study; ravulizumab; respiratory distress syndrome, adult; Ultomiris; viral
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Pneumonia, Viral; COVID-19; Pneumonia; Severe Acute Respiratory Syndrome | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Ravulizumab + BSC (Experimental)
  Interventions: Biological: Ravulizumab; Other: BSC
- Group 2 - BSC alone (Other)
  Interventions: Other: BSC

INTERVENTIONS:
Biological: Ravulizumab — Weight-based doses of ravulizumab were administered intravenously on Days 1, 5, 10, and 15.
  Other Names: Ultomiris; ALXN1210
  Arms: Group 1 - Ravulizumab + BSC
Other: BSC — Participants received medications, therapies, and interventions per standard hospital treatment protocols.

SUMMARY:
This study evaluated the efficacy, safety, pharmacokinetics, and pharmacodynamics of ravulizumab administered in adult participants with coronavirus disease 2019 (COVID-19) severe pneumonia, acute lung injury, or acute respiratory distress syndrome. Participants were randomly assigned to receive ravulizumab in addition to best supportive care (BSC) (2/3 of the participants) or BSC alone (1/3 of the participants). BSC consisted of medical treatment and/or medical interventions per routine hospital practice.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female participants ≥ 18 years of age and ≥ 40 kilograms at the time of providing informed consent.
2. Confirmed diagnosis of severe acute respiratory syndrome coronavirus 2 infection (for example, via polymerase chain reaction and/or antibody test) presenting as severe COVID-19 requiring hospitalization.
3. Severe pneumonia, acute lung injury, or acute respiratory distress syndrome confirmed by computed tomography or X-ray at Screening or within the 3 days prior to Screening, as part of the participant's routine clinical care.
4. Respiratory distress requiring mechanical ventilation, which can be either invasive (requiring endotracheal intubation) or noninvasive (with continuous positive airway pressure or bilevel positive airway pressure).
5. Female participants of childbearing potential and male participants with female partners of childbearing potential must follow protocol specified contraception guidance for avoiding pregnancy for 8 months after treatment with the study drug.

Exclusion Criteria:

1. Participant was not expected to survive for more than 24 hours.
2. Participant was on invasive mechanical ventilation with intubation for more than 48 hours prior to Screening.
3. Severe pre-existing cardiac disease (that is, New York Heart Association Class 3 or Class 4, acute coronary syndrome or persistent ventricular tachyarrhythmias).
4. Participant had an unresolved Neisseria meningitidis infection.
5. Used the following medications and therapies:

   * Current treatment with a complement inhibitor or
   * Intravenous immunoglobulin within 4 weeks prior to randomization on Day 1
6. Treatment with investigational therapy in a clinical study within 30 days before randomization, or within 5 half-lives of that investigational therapy, whichever was greater. Exceptions:

   * Investigational therapies were allowed if received as part of BSC through an expanded access protocol or emergency approval for the treatment of COVID-19.
   * Investigational antiviral therapies (such as remdesivir) were allowed even if received as part of a clinical study.
7. Female participants who were breastfeeding or who have a positive pregnancy test result at Screening.
8. History of hypersensitivity to any ingredient contained in the study drug, including hypersensitivity to murine proteins.
9. Participant who was not currently vaccinated against Neisseria meningitidis, unless the participant agrees to receive prophylactic treatment with appropriate antibiotics for at least 8 months after the last infusion of study drug or until at least 2 weeks after the participant receives vaccination against Neisseria meningitidis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (24):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - LAC/USC Health Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Health System, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Mayo Clinic Health System in Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System, La Crosse, Wisconsin
- France (3):
  - Hôpital Raymond Poincaré, Garches, Hauts De Seine
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
- Japan (3):
  - Jikei University Hospital, Minato-Ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City, Tokyo-To
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
- United Kingdom (5):
  - King's College Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - St James's University Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] WHO. Clinical management of severe acute respiratory infection when novel coronavirus (2019-nCoV) infection is suspected. Interim guidance, 28 January 2020.
- [Result] McEneny-King AC, Monteleone JPR, Kazani SD, Ortiz SR. Pharmacokinetic and Pharmacodynamic Evaluation of Ravulizumab in Adults with Severe Coronavirus Disease 2019. Infect Dis Ther. 2021 Jun;10(2):1045-1054. doi: 10.1007/s40121-021-00425-7. Epub 2021 Apr 7. PMID 33826106
- [Result] Smith K, Pace A, Ortiz S, Kazani S, Rottinghaus S. A Phase 3 Open-label, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Intravenously Administered Ravulizumab Compared with Best Supportive Care in Patients with COVID-19 Severe Pneumonia, Acute Lung Injury, or Acute Respiratory Distress Syndrome: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jul 13;21(1):639. doi: 10.1186/s13063-020-04548-z. PMID 32660611
- [Derived] Annane D, Pittock SJ, Kulkarni HS, Pickering BW, Khoshnevis MR, Siegel JL, Powell CA, Castro P, Fujii T, Dunn D, Smith K, Mitter S, Kazani S, Kulasekararaj A. Intravenous ravulizumab in mechanically ventilated patients hospitalised with severe COVID-19: a phase 3, multicentre, open-label, randomised controlled trial. Lancet Respir Med. 2023 Dec;11(12):1051-1063. doi: 10.1016/S2213-2600(23)00082-6. Epub 2023 Mar 20. PMID 36958364
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Java A, Apicelli AJ, Liszewski MK, Coler-Reilly A, Atkinson JP, Kim AH, Kulkarni HS. The complement system in COVID-19: friend and foe? JCI Insight. 2020 Aug 6;5(15):e140711. doi: 10.1172/jci.insight.140711. PMID 32554923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 210 participants screened, 8 (3.8%) participants were screen failures. A total of 202 participants were randomized and treated.
Groups:
- Group 1 - Ravulizumab + BSC: Ravulizumab: Weight-based doses of ravulizumab were administered intravenously on Days 1, 5, 10, and 15. BSC: Participants received medications, therapies, and interventions per standard hospital treatment protocols.
- Group 2 - BSC Alone: Participants received medications, therapies, and interventions per standard hospital treatment protocols
Period: Overall Study
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Started | 135 | 67
Intent to Treat (ITT) Population (The ITT Population consisted of all randomized participants. Participants were analyzed as randomized.) | 135 | 66
Pharmacokinetic (PK) (The PK Set included participants in the ITT population with at least one postdose PK result.) | 127 | 52
Safety Population (All randomized participants who received at least 1 dose of study drug. Participants were analyzed as treated.) | 127 | 67
Completed | 125 | 58
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Did Not Meet Inclusion/Exclusion Criteria | 2 | 0
Not completed — Not Qualified due to History of Anaphylaxis | 1 | 0
Not completed — Unable to Provide Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: The ITT Population consisted of all randomized participants. Participants were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone | Total
Number analyzed (Participants) | 135 | 66 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (13.23) | 63.5 (12.40) | 63.3 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 23 | 62
  Male | 96 | 43 | 139
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 100 | 46 | 146
  Hispanic or Latino | 27 | 11 | 38
  Missing/Unknown | 7 | 5 | 12
  Not reported | 1 | 4 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 72 | 40 | 112
  Black or African American | 20 | 7 | 27
  Missing/Unknown | 17 | 5 | 22
  Other | 13 | 5 | 18
  Asian | 9 | 6 | 15
  Not Reported | 4 | 2 | 6
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Survival (Based On All-Cause Mortality) in Participants in the ITT Population At Day 29
Description: Survival (based on all-cause mortality) in Participants in the ITT Population at Day 29 was analyzed. The result for the survival was estimated survival combined over all imputations.
Time Frame: Day 29
Population: The ITT Population consisted of all randomized participants. Participants were analyzed as randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 135 | 66
Percentage of participants | 57.6 | 59.7
Statistical Analysis 1: Comparison: Group 1 - Ravulizumab + BSC vs Group 2 - BSC Alone; Test type: Other; p = 0.6059, Mantel Haenszel — One-sided Mantel-Haenszel test of the difference in two proportions stratified by intubated or not intubated on Day 1 and a family-wise Type I error of 0.025; Risk Difference (RD) = -0.0205, 95% CI 2-sided [-0.1703 to 0.1293] — Two-sided 95% confidence interval using the Sato variance estimator, combined overall imputations

2. Secondary Outcome: Number Of Days Free Of Mechanical Ventilation At Day 29
Description: The number of days free of mechanical ventilation was defined as the total number of days from Day 1 to Day 29 without invasive or non-invasive mechanical ventilation.
Time Frame: Day 29
Population: The ITT Population consisted of all randomized participants. Participants were analyzed as randomized. Here, 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 129 | 62
Days | 6.79 [4.79 to 8.80] | 6.81 [4.19 to 9.43]

3. Secondary Outcome: Number of Days the Participants Were Alive and Not in ICU
Description: The number of days that the participants were alive and not in the ICU from Day 1 through Day 29 are presented.
Time Frame: Day 1 through Day 29
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 129 | 62
Days | 6.09 [4.31 to 7.87] | 6.71 [4.38 to 9.03]

4. Secondary Outcome: Change From Baseline In Sequential Organ Failure Assessment (SOFA) At Day 29
Description: Baseline was defined as the last available assessment on or before Day 1 for all participants. Participants were evaluated using the SOFA score, an assessment tool that included a review of 6 organ systems: respiratory, renal, hepatic, cardiac, coagulation, and central nervous system. Each organ system was scored from 0 to 4 points using the worst value observed within the previous 24 hours. The total score ranged from 0 to 24, with a higher score indicating a worse condition.
Time Frame: Baseline, Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 42 | 17
Units on a scale | -2.0 (6.25) | -4.5 (4.90)

5. Secondary Outcome: Change From Baseline In Peripheral Capillary Oxygen Saturation/Fraction Of Inspired Oxygen (SpO2/FiO2) At Day 29
Description: Oxygenation was measured using the SpO2 and the amount of supplemental oxygen as measured by the FiO2 received by taking the ratio of these 2 measures at the same time point.
Time Frame: Baseline, Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 38 | 17
ratio | 62.5 (112.43) | 134.0 (104.35)

6. Secondary Outcome: Number of Days the Participants Were Alive and Not in the Hospital
Description: The number of days that the participants were alive and not in the hospital from Day 1 through Day 29 are presented.
Time Frame: Day 1 through Day 29
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 129 | 62
Days | 3.02 [1.76 to 4.29] | 3.47 [1.83 to 5.12]

7. Secondary Outcome: Estimated Number of Participants Alive At Up To Day 60 and At Up To Day 90
Description: For this analysis, 2 participants in Group 1 (Ravulizumab + BSC) and 1 participant in Group 2 (BSC Alone) were censored at Day 90. The estimated number of participants alive for this analysis was calculated using the method of Kaplan and Meier (KM) and compared using a log-rank test stratified by intubated or not intubated on Day 1 as a sensitivity analysis. This Outcome Measure was designed to project an estimate of how many participants would be alive and not the actual number of alive participants. All-Cause Mortality data is provided in the Adverse Events Section.
Time Frame: Up to Day 60 and Up to Day 90
Population: The ITT Population consisted of all randomized participants. Participants were analyzed as randomized. Here, "Number Analyzed" signifies those participants who were evaluable for the assessment at the specified time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 135 | 66
Participants
  Day 60 | 60 | 29
  Day 90: number analyzed (Participants) | 133 | 65
  Day 90 | 49 | 20

8. Secondary Outcome: Serum Ravulizumab Concentrations Prior to Dosing on Day 1 and Day 29
Description: Results are reported in micrograms/milliliter (μg/mL).
Time Frame: Day 1 and Day 29
Population: Pharmacokinetics/Pharmacodynamics (PK/PD) Population: participants in the ITT population with at least 1 postdose PK or PD result.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group 1 - Ravulizumab + BSC
Number analyzed (Participants) | 126
μg/mL
  Day 1 (predose): number analyzed (Participants) | 116
  Day 1 (predose) | 0.00 (0.00)
  Day 29 (predose): number analyzed (Participants) | 44
  Day 29 (predose) | 231.35 (149.741)

9. Secondary Outcome: Change From Baseline In Serum Free Complement Component 5 Concentrations At Day 29
Time Frame: Baseline, Day 29
Population: PK/PD Population: participants in the ITT population with at least 1 postdose PK or PD result. Here, 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 43 | 14
μg/mL | -156.31 (61.599) | 21.79 (67.918)

10. Secondary Outcome: Change From Baseline In Terminal Complement Complex C5b-9 At Day 29
Time Frame: Baseline, Day 29
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
Number analyzed (Participants) | 43 | 14
ug/L | -133.23 (202.070) | -277.21 (604.742)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 90
Description: Data for All-Cause Mortality was collected for the ITT Population (all randomized participants; participants were analyzed as randomized). Serious and Other (Not Including Serious) Adverse Events were collected for the Safety Population (all randomized participants who received at least 1 dose of study drug; participants were analyzed as treated).
Arm/Group | Group 1 - Ravulizumab + BSC | Group 2 - BSC Alone
All-Cause Mortality (participants affected / at risk) | 55/135 | 25/66
Serious Adverse Events (participants affected / at risk) | 79/127 | 38/67
Other Adverse Events (participants affected / at risk) | 97/127 | 49/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Ravulizumab + BSC (N=127) | Group 2 - BSC Alone (N=67)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 14 (14) | 6 (6)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 13 (15) | 3 (5)
COVID-19 pneumonia (Infections and infestations) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (3) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Systemic candida (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood beta-D-glucan positive (Investigations) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Shock hemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Ravulizumab + BSC (N=127) | Group 2 - BSC Alone (N=67)
Hypotension (Vascular disorders) | 16 (18) | 8 (10)
Anaemia (Blood and lymphatic system disorders) | 13 (15) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 12 (12) | 5 (5)
Pyrexia (General disorders) | 10 (12) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 14 (14) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 9 (10) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (9) | 6 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 11 (11) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (4)
Hypertension (Vascular disorders) | 9 (9) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 7 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (6)
Bradycardia (Cardiac disorders) | 6 (6) | 4 (4)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)

LIMITATIONS AND CAVEATS:
Enrollment of participants was paused on 13-Jan-2021. At that time, 202 participants had been randomized. An interim analysis for efficacy and futility was conducted on data from the first 122 participants who completed the Primary Evaluation Period. The analysis showed that the study met the prespecified stopping criteria for futility. After review of all participant data, Alexion terminated the study on 01-Sep-2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT04369469/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT04369469/SAP_001.pdf